CLINICAL TRIAL: NCT05889325
Title: Efficacy and Safety of Irinotecan-eluting HepaSphere Transarterial Chemoembolization Combined With Hepatic Arterial Infusion Chemotherapy for Unresectable Colorectal Liver Metastases
Brief Title: To Evaluate the Performance of HepaSphere Transarterial Chemoembolization Combined With Hepatic Arterial Infusion Chemotherapy on Unresectable Colorectal Liver Metastases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Other Study IDs: CRCLM-HEPA-HAIC-001
Record Dates: First submitted 2023-05-08; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Colorectal Liver Metastases (CRCLM)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: DEB-TACE plus HAIC — the patients received HepaSphere DEB-TACE plus HAIC

SUMMARY:
Both drug-eluting bead transarterial chemoembolization (DEB-TACE) and hepatic arterial infusion chemotherapy (HAIC) are recommended for unresectable colorectal liver metastases (CRLM) treatment. However, the combined application of DEB-TACE and HAIC is not widely accepted. The aim of this single-center retrospective study was to evaluate the efficacy and safety of Irinotecan-eluting HepaSphere chemoembolization combined with HAIC for unresectable CRLM

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years old
* Gender: no limitation
* Histologically or cytologically documented advanced colorectal carcinoma with unresectable liver metastasis (existence of extrahepatic metastasis is acceptable)
* Subjects must have at least one measurable lesion per RECIST v1.1
* Patients only received treatment with HepaSphere combined with hepatocellular arterial infusion chemotherapy (HAIC) as interventional therapy during the observation period
* Child-Pugh: A-B
* ECOG: 0-2.

Exclusion Criteria:

* Other malignant tumors in the past 5 years
* Drug-eluting beads from other manufacturers were used during DEB-TACE
* DEB-TACE combined with HAIC was used as postoperative adjuvant therapy
* Pre- or post-surgery relevant examination results were unavailable
* Imaging information for effectiveness evaluation was unavailable
* Follow-up failure due to patient information errors, loss, refusal, etc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a retrospective observation study. All of the patients included in this study were diagnosed as advanced colorectal carcinoma with unresectable liver metastasis. In additional, they received only HepaSphere DEB-TACE plus HAIC as the interventional therapy in a period of time from 2018 to 2022 . There is no any intervention in this study
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 3 years
  Progression-free survival is defined as the time from the start of treatment HepaSphere DEB-TACE plus HAIC until the first documentation of disease progression or death due to any cause, whichever occurs first

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 3 years
  Overall survival is defined as the time from the start of treatment with HepaSphere DEB-TACE plus HAIC until death due to any cause
Objective Response Rate (ORR) | Up to 3 years
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1
Duration of Response (DoR) | Up to 3 years
  Duration of response is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No